CLINICAL TRIAL: NCT03187834
Title: Antibiotic Resistance and Microbiome in Children Aged 6-59 Months in Nouna, Burkina Faso
Acronym: ARMCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-22036
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Child Development
Keywords: infection; azithromycin; amoxicillin; co-trimoxazole; trachoma; mass treatment
MeSH Terms: conditions — Infections; Trachoma | interventions — Azithromycin; Amoxicillin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Households will be randomized to one of four treatment arms (azithromycin, cotrimoxazole, amoxicillin, or placebo), and each child age 6-59 months in the household will receive 5 days of treatment. One child within each of the antibiotic households will be randomly selected to receive placebo instead of the antibiotc, to allow for study of indirect effects of antibiotic use
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Azithromycin (Active Comparator): Comparison of nasopharyngeal and rectal microbiome in children receiving Azithromycin versus children receiving placebo Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm and treated for 5 days.
  Children will receive treatment everyday, once a day as is:
  Azithromycin: 10 mg/kg once daily on Day 1, then 5 mg/kg once daily Days 2-5
  Interventions: Drug: Azithromycin
- Amoxicillin (Active Comparator): Comparison of nasopharyngeal and rectal microbiome in children receiving Amoxicillin versus children receiving placebo Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm.
  Children will receive treatment everyday, twice a day as is:
  Amoxicillin: 25 mg/kg/day, divided into twice daily doses for Days 1-5
  Interventions: Drug: Amoxicillin
- Cotrimoxazole (Active Comparator): Comparison of nasopharyngeal and rectal microbiome in children receiving Cotri-moxazole versus children receiving placebo Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm.
  Children will receive treatment everyday, once a day as is:
  Co-trimoxazole: 240 mg daily for Days 1-5
  Interventions: Drug: Cotrimoxazole
- Placebo (Placebo Comparator): Comparison of nasopharyngeal and rectal microbiome in children receiving placebo versus children receiving antibiotics Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm.
  Children will receive Placebo everyday, once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Children in this arm will receive Azithromycin once a day.
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Amoxicillin — Children in this arm will receive Amoxicillin twice a day.
  Arms: Amoxicillin
Drug: Cotrimoxazole — Children in this arm will receive co-trimoxazole once a day.
  Arms: Cotrimoxazole
Drug: Placebo — Children in this arm will receive Placebo once a day.
  Arms: Placebo

SUMMARY:
The use of antibiotics has saved millions of human lives, however consumption of antibiotics can select for antibiotic resistant organisms and may lead to changes in commensal microbiome. This study is designed to estimate the effect of antibiotic consumption on microbiome in a rural region of rural Burkina Faso. Changes in the intestinal and nasopharyngeal microbiome and resistome following a short course of antibiotics will be measured.

DETAILED DESCRIPTION:
This study is designed to better understand the effect of a short course of antibiotics on changes in intestinal and nasopharyngeal microbiome on treated children and untreated household contacts. The investigators hypothesize that a short course of antibiotics will lead to decreased bacterial diversity shortly after completion of the antibiotic course, and higher probability of identification of bacterial resistance genes in rectal and nasopharyngeal samples. The investigators hypothesize that a 5-day course of antibiotics (azithromycin, amoxicillin, or co-trimoxazole) will lead to significantly decreased intestinal and nasopharyngeal bacterial diversity among children aged 6-59 months.

Specific Aim 1. Determine the effect of treatment with antibiotics on microbiome diversity in children aged 6-59 months following a 5-day course of antibiotics.

Specific Aim 1A. Determine the direct effect of a 5-day course of azithromycin, amoxicillin, or co-trimoxazole on intestinal and nasopharyngeal bacterial diversity in children aged 6-59 months compared to no treatment.

Specific Aim 1B. Determine the indirect effect of antibiotic treatment of children in a household on intestinal and nasopharyngeal bacterial diversity in an untreated child aged 6-59 months.

Specific Aim 1C. Assess the association between intestinal bacterial diversity and anthropometry in a population-based sample of children.

ELIGIBILITY:
Inclusion Criteria:

* Households will be eligible for inclusion in the study if they have 2 or more children aged 6 months to 59 months currently residing in the household. Children from the household will be eligible if they are 6-59 months of age and are not currently receiving antibiotic treatment

Exclusion Criteria:

* Children who are allergic to any of the study antibiotics will be excluded. Individuals aged under 6 months and 5 years or older will be excluded. Children already receiving antibiotics for an ongoing disease will be excluded.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Lietman, MD, Principal Investigator — UCSF F.I. Proctor Foundation; Catherine E Oldenburg, ScD, Study Director — UCSF F.I. Proctor Foundation
Locations (2):
- UCSF Proctor Foundation, San Francisco, California, United States
- Centre de Recherche en Santé de Nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldenburg CE, Hinterwirth A, Worden L, Sie A, Dah C, Ouermi L, Coulibaly B, Zhong L, Chen C, Ruder K, Lietman TM, Keenan JD, Doan T. Indirect effect of oral azithromycin on the gut resistome of untreated children: a randomized controlled trial. Int Health. 2021 Feb 24;13(2):130-134. doi: 10.1093/inthealth/ihaa029. PMID 32556194
- [Derived] Dennis EG, Sie A, Ouermi L, Dah C, Tapsoba C, Zabre P, Barnighausen T, O'Brien KS, Lebas E, Keenan JD, Oldenburg CE. Short-term weight gain among preschool children in rural Burkina Faso: a secondary analysis of a randomised controlled trial. BMJ Open. 2019 Jul 29;9(7):e029634. doi: 10.1136/bmjopen-2019-029634. PMID 31362969
- [Derived] Oldenburg CE, Sie A, Coulibaly B, Ouermi L, Dah C, Tapsoba C, Barnighausen T, Lebas E, Arzika AM, Cummings S, Zhong L, Lietman TM, Keenan JD, Doan T. Indirect Effect of Azithromycin Use on the Intestinal Microbiome Diversity of Untreated Children: A Randomized Trial. Open Forum Infect Dis. 2019 Feb 6;6(3):ofz061. doi: 10.1093/ofid/ofz061. eCollection 2019 Mar. PMID 30895203
- [Derived] Oldenburg CE, Sie A, Coulibaly B, Ouermi L, Dah C, Tapsoba C, Barnighausen T, Ray KJ, Zhong L, Cummings S, Lebas E, Lietman TM, Keenan JD, Doan T. Effect of Commonly Used Pediatric Antibiotics on Gut Microbial Diversity in Preschool Children in Burkina Faso: A Randomized Clinical Trial. Open Forum Infect Dis. 2018 Nov 2;5(11):ofy289. doi: 10.1093/ofid/ofy289. eCollection 2018 Nov. PMID 30515431
- [Derived] Sie A, Dah C, Ouermi L, Tapsoba C, Zabre P, Barnighausen T, Lebas E, Arzika AM, Snyder BM, Porco TC, Lietman TM, Keenan JD, Oldenburg CE. Effect of Antibiotics on Short-Term Growth among Children in Burkina Faso: A Randomized Trial. Am J Trop Med Hyg. 2018 Sep;99(3):789-796. doi: 10.4269/ajtmh.18-0342. Epub 2018 Jul 12. PMID 30014828

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: household
Groups:
- Amoxicillin Households: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, twice a day as is:
  Amoxicillin: 25 mg/kg/day, divided into twice daily doses for Days 1-5
  Amoxicillin Households - Antibiotic: Children in this arm will receive Amoxicillin twice a day.
- Azithromycin Households: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Azithromycin: 10 mg/kg once daily on Day 1, then 5 mg/kg once daily Days 2-5
  Azithromycin Households - Antibiotic: Children in this arm will receive Azithromycin once a day.
- Cotrimoxazole Households: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Co-trimoxazole: 240 mg daily for Days 1-5
  Cotrimoxazole: Children in this arm will receive co-trimoxazole once a day.
- Placebo: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo. In placebo households, both children received placebo.
Period: Overall Study
Arm/Group | Amoxicillin Households | Azithromycin Households | Cotrimoxazole Households | Placebo
Started | 62; 31 household | 62; 31 household | 62; 31 household | 62; 31 household
Receive Antibiotic | 31; 31 household | 31; 31 household | 31; 31 household | 31; 31 household
Receive Placebo | 31; 31 household | 31; 31 household | 31; 31 household | 31; 31 household
Completed | 57; 30 household | 58; 31 household | 56; 31 household | 58; 31 household
Not Completed | 5; 1 household | 4; 0 household | 6; 0 household | 4; 0 household
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2
Not completed — Had invalid anthropometric measurements | 5 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Children between 6 and 59 months of age and with parental consent. Data were only collected from children. In each arm, one children was given Antibiotic and one children was given Placebo. The baseline characteristics were reported separately in analysis and papers.
Groups:
- Amoxicillin Households - Antibiotic: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, twice a day as is:
  Amoxicillin: 25 mg/kg/day, divided into twice daily doses for Days 1-5
  Amoxicillin Households - Antibiotic: Children in this arm will receive Amoxicillin twice a day.
- Amoxicillin Households - Placebo: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Amoxicillin Households - Placebo: Children in this arm will receive Placebo.
- Azithromycin Households - Antibiotic: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Azithromycin: 10 mg/kg once daily on Day 1, then 5 mg/kg once daily Days 2-5
  Azithromycin Households - Antibiotic: Children in this arm will receive Azithromycin once a day.
- Azithromycin Households - Placebo: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Azithromycin Households - Placebo: Children in this arm will receive Placebo.
- Cotrimoxazole Households - Antibiotic: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Co-trimoxazole: 240 mg daily for Days 1-5
  Cotrimoxazole: Children in this arm will receive co-trimoxazole once a day.
- Cotrimoxazole Households - Placebo: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Cotrimoxazole Households - Placebo: Children in this arm will receive Placebo.
- Total: Total of all reporting groups
Arm/Group | Amoxicillin Households - Antibiotic | Amoxicillin Households - Placebo | Azithromycin Households - Antibiotic | Azithromycin Households - Placebo | Cotrimoxazole Households - Antibiotic | Cotrimoxazole Households - Placebo | Placebo | Total
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 62 | 248
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 35 [23 to 52] | 36 [26 to 53] | 29 [21 to 51] | 42 [30 to 47] | 37 [23 to 48] | 40 [23 to 50] | 38 [30 to 49] | 37 [25 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 18 | 12 | 20 | 19 | 24 | 125
  Male | 17 | 13 | 13 | 19 | 11 | 12 | 38 | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Wasted [Count of Participants; unit: Participants] — Defined as Weight-for-height Z-score (WHZ) < -2 SD.
  Participants | 2 | 3 | 2 | 3 | 2 | 7 | 6 | 25
Stunted [Count of Participants; unit: Participants] — Defined as Height-for-age Z-score (HAZ) < -2 SD.
  Participants | 8 | 7 | 8 | 7 | 4 | 11 | 7 | 52
Underweight [Count of Participants; unit: Participants] — Defined as Weight-for-age Z-score (WAZ) < -2 SD.
  Participants | 5 | 3 | 4 | 4 | 3 | 10 | 6 | 35
Visited healthcare facility in past 30 days [Count of Participants; unit: Participants] | 6 | 2 | 4 | 2 | 6 | 8 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Simpson's Index of Diversity (Alpha Diversity) in Intestinal Microbiome
Description: The primary outcome of the study was pre-specified as α-diversity (inverse Simpson's) at the genus level, expressed in effective number. Simpson's Alpha Diversity were obtained at Baseline and Post-treatment in this study. The minimum of Simpson's index of diversity is 0, there is no maximum. Higher Simpson's index of diversity means more diverse. There are no subscales.
Time Frame: Baseline and Day 9
Population: 248 children in 124 households were enrolled and randomized to 1 of the 3 antibiotic regimens or placebo. Of these, 124 children were randomized within their household to receive treatment and are included in this analysis. Of these children, 9 children were lost to follow-up.
  The samples from Amoxicillin Households - Placebo, Azithromycin Households - Placebo, Cotrimoxazole Households - Placebo and half of placebo (31 participants) were not collected and analyzed, due to limited budget.
Measure: Mean (95% Confidence Interval); unit: Index score
Groups:
- Amoxicillin: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, twice a day as is:
  Amoxicillin: 25 mg/kg/day, divided into twice daily doses for Days 1-5 Amoxicillin Households - Antibiotic: Children in this arm will receive Amoxicillin twice a day.
- Azithromycin: Comparison of nasopharyngeal and rectal microbiome in children receiving Azithromycin versus children receiving placebo Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm and treated for 5 days.
  Children will receive treatment everyday, once a day as is:
  Azithromycin: 10 mg/kg once daily on Day 1, then 5 mg/kg once daily Days 2-5
  Azithromycin: Children in this arm will receive Azithromycin once a day.
- Cotrimoxazole: Comparison of nasopharyngeal and rectal microbiome in children receiving Cotri-moxazole versus children receiving placebo Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm.
  Children will receive treatment everyday, once a day as is:
  Co-trimoxazole: 240 mg daily for Days 1-5
  Cotrimoxazole: Children in this arm will receive co-trimoxazole once a day.
- Placebo: Comparison of nasopharyngeal and rectal microbiome in children receiving placebo versus children receiving antibiotics Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm.
  Children will receive Placebo everyday, once a day.
  Placebo: Children in this arm will receive Placebo once a day.
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 31 | 31 | 31 | 31
Index score
  Baseline | 10.2 [8.8 to 11.5] | 8.8 [7.5 to 10.1] | 9.7 [8.2 to 11.2] | 9.6 [8.6 to 10.7]
  Post-treatment: number analyzed (Participants) | 27 | 30 | 29 | 29
  Post-treatment | 8.3 [7.0 to 9.6] | 6.6 [5.5 to 7.8] | 8.3 [6.9 to 9.7] | 9.8 [8.7 to 10.9]

2. Secondary Outcome: Simpson's Index of Diversity (Alpha Diversity) in Microbiome
Description: Direct and indirect effect of antibiotics on alpha diversity from rectal samples
Time Frame: Day 9
Population: rectal samples were not analyzed due to limited budget - samples were collected but not analyzed and never will be analyzed
Arm/Group | Amoxicillin Households | Azithromycin Households | Cotrimoxazole Households | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Weight-for-height Z-score
Description: Nutritional status as determined by weight-for-height Z-score vs. Placebo household Weight-for-height Z-score in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Weight-for-height Z (WHZ) scores were calculated based on the 2006 World Health Organization (WHO) standards. The mean of the 2006 population standards is 0. Lower standard deviations = worse outcomes. A cutoff of < -2 means moderately wasted (WHZ). A cutoff of < -3 means wasted (WHZ).
Time Frame: Day 35
Population: In Amoxicillin, Azithromycin, Cotrimoxazole households, children assigned to receive antibiotic and placebo were analyzed separately, showed in different row below.
Measure: Mean (Standard Deviation); unit: z score
Groups:
- Azithromycin: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Azithromycin: 10 mg/kg once daily on Day 1, then 5 mg/kg once daily Days 2-5 Azithromycin Households - Antibiotic: Children in this arm will receive Azithromycin once a day.
- Cotrimoxazole: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Co-trimoxazole: 240 mg daily for Days 1-5 Cotrimoxazole: Children in this arm will receive co-trimoxazole once a day.
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 57 | 58 | 56 | 58
z score
  Children who received Antibiotic: number analyzed (Participants) | 29 | 29 | 29 | 0
  Children who received Antibiotic | -0.24 (0.92) | -0.71 (0.98) | -0.27 (0.91) |
  Children who received Placebo: number analyzed (Participants) | 28 | 29 | 27 | 58
  Children who received Placebo | -0.52 (1.05) | -0.17 (0.85) | -0.49 (1.11) | -0.28 (1.00)

4. Secondary Outcome: Height-for-age Z-score
Description: Nutritional status as determined by height-for-age Z-score Height-for-age Z-score in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Height-for-age Z (HAZ) score were calculated based on the 2006 World Health Organization (WHO) standards. The mean of the 2006 population standards is 0. Lower standard deviations = worse outcomes. A cutoff of < -2 means moderately stunted (HAZ). A cutoff of < -3 means severely stunted (HAZ).
Time Frame: Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 57 | 58 | 56 | 58
z score
  Children who received Antibiotic: number analyzed (Participants) | 29 | 29 | 29 | 0
  Children who received Antibiotic | -0.80 (1.19) | -0.92 (1.13) | -0.69 (1.00) |
  Children who received Placebo: number analyzed (Participants) | 28 | 29 | 27 | 58
  Children who received Placebo | -0.73 (1.11) | -1.16 (1.34) | -1.38 (0.94) | -0.59 (1.08)

5. Secondary Outcome: Weight-for-age Z-score
Description: Nutritional status as determined by weight-for-age Z-score vs. Placebo household Weight-for-age Z-score in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Weight-for-age Z-score (WAZ) scores were calculated based on the 2006 World Health Organization (WHO) standards. The mean of the 2006 population standards is 0. Lower standard deviations = worse outcomes. A cutoff of < -2 means moderately underweight (WAZ). A cutoff of < -3 means severely underweight (WAZ).
Time Frame: Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 57 | 58 | 56 | 58
Z score
  Children who received Antibiotic: number analyzed (Participants) | 29 | 29 | 29 | 0
  Children who received Antibiotic | -0.60 (0.87) | -1.01 (0.95) | -0.58 (0.94) |
  Children who received Placebo: number analyzed (Participants) | 28 | 29 | 27 | 58
  Children who received Placebo | -0.78 (0.89) | -0.78 (1.02) | -1.12 (1.04) | -0.53 (0.97)

6. Secondary Outcome: Mid-upper Arm Circumference
Description: Nutritional status as determined by mid-upper arm circumference in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Mid-upper arm circumference (MUAC) in each antibiotic group compared with placebo 4 weeks after last antibiotic dose.
  MUAC is a measure to assess nutritional status. It is measured on a straight left arm, mid-way between the tip of the shoulder and the tip of the elbow. It identifies acute malnutrition and is commonly used in children 6-59 months of age as well as pregnant women. MUAC less than 115 mm indicates severe wasting or severe acute malnutrition (SAM). MUAC greater than or equal to 115 mm and less than 125 mm indicates moderate wasting or moderate acute malnutrition (MAM).
Time Frame: Day 35
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 57 | 58 | 56 | 58
mm
  Children who received Antibiotic: number analyzed (Participants) | 29 | 29 | 29 | 0
  Children who received Antibiotic | 15.01 (0.92) | 14.53 (1.11) | 15.49 (0.98) |
  Children who received Placebo: number analyzed (Participants) | 28 | 29 | 27 | 58
  Children who received Placebo | 14.90 (1.10) | 15.15 (1.01) | 14.83 (1.36) | 15.23 (1.23)

7. Secondary Outcome: Shannon's Index of Diversity (Alpha Diversity) in Intestinal Microbiome
Description: Shannon's Alpha Diversity at Baseline and Post-treatment. combines richness and diversity. Shannon's index of diversity (alpha diversity) measures both the number of species and the inequality between species abundances. A large value is given by the presence of many species with well balanced abundances.
Time Frame: Baseline and Day 9 (Post- Treatment)
Population: 248 children in 124 households were enrolled and randomized to 1 of the 3 antibiotic regimens or placebo. Of these, 124 children were randomized within their household to receive treatment and are included in this analysis. Of these children, 9 children were lost to follow-up.
  The samples for children who received placebo in Amoxicillin Households, Azithromycin Households, Cotrimoxazole Households and half of placebo (31 participants) were not collected and analyzed, due to limited budget.
Measure: Mean (95% Confidence Interval); unit: Index score
Groups:
- Amoxicillin: Comparison of nasopharyngeal and rectal microbiome in children receiving Amoxicillin versus children receiving placebo Children aged 6 months to 59 months will be measured and weighed then, they will be randomized to one of the study arm.
  Children will receive treatment everyday, twice a day as is:
  Amoxicillin: 25 mg/kg/day, divided into twice daily doses for Days 1-5
  Amoxicillin: Children in this arm will receive Amoxicillin twice a day.
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 31 | 31 | 31 | 31
Index score
  Baseline | 16.6 [14.5 to 18.7] | 14.6 [13.0 to 16.2] | 15.6 [13.4 to 17.8] | 15.4 [14.1 to 16.7]
  Post-treatment: number analyzed (Participants) | 27 | 30 | 29 | 29
  Post-treatment | 13.9 [12.1 to 15.8] | 11.0 [9.3 to 12.7] | 13.5 [11.6 to 15.4] | 16.0 [14.3 to 17.8]

8. Secondary Outcome: Shannon's Index of Diversity (Alpha Diversity) in Nasopharyngeal Microbiome
Description: Direct and indirect effects of antibiotics on Shannon's index of bacterial diversity
Time Frame: Day 9
Population: Nasopharyngeal samples were not analyzed, due to limited budget - samples were collected but not analyzed and never will be analyzed
Arm/Group | Amoxicillin Households | Azithromycin Households | Cotrimoxazole Households | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: L1-norm Distance on Bacterial Reads (Intestinal)
Description: L1-norm distance on bacterial reads (intestinal) - L1 norm is equivalent to Shannon's diversity. Shannon's Alpha Diversity combines richness and diversity. Shannon's index of diversity (alpha diversity) measures both the number of species and the inequality between species abundances. A large value is given by the presence of many species with well balanced abundances.
Time Frame: Baseline and Day 9 (Post- Treatment)
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: Index score
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 31 | 31 | 31 | 31
Index score
  Baseline | 16.6 [14.5 to 18.7] | 14.6 [13.0 to 16.2] | 15.6 [13.4 to 17.8] | 15.4 [14.1 to 16.7]
  Post-treatment: number analyzed (Participants) | 27 | 30 | 29 | 29
  Post-treatment | 13.9 [12.1 to 15.8] | 11.0 [9.3 to 12.7] | 13.5 [11.6 to 15.4] | 16.0 [14.3 to 17.8]

10. Secondary Outcome: L1-norm Distance on Bacterial Reads (Nasopharyngeal)
Description: L1-norm distance on bacterial reads (nasopharyngeal)
Time Frame: Day 9
Population: Nasopharyngeal samples were not analyzed due to limited budget- samples were collected but not analyzed and never will be analyzed
Arm/Group | Amoxicillin Households | Azithromycin Households | Cotrimoxazole Households | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: L2-norm Distance on Bacterial Reads (Intestinal)
Description: L2-norm distance on bacterial reads (intestinal) - L2 norm is equivalent to Simpson's diversity. Simpson's Alpha Diversity were obtained at Baseline and Post-treatment in this study. The minimum of Simpson's index of diversity is 0, there is no maximum. Higher Simpson's index of diversity means more diverse. There are no subscales.
Time Frame: Baseline and Day 9 (Post- Treatment)
Population: 248 children in 124 households were enrolled and randomized to 1 of the 3 antibiotic regimens or placebo. Of these, 124 children were randomized within their household to receive treatment and are included in this analysis. Of these children, 9 children were lost to follow-up.
  Indirect effect (antibiotic household - placebo) was not analyzed. we will not analyzed these biological specimens because no funding are available for this. Only direct effect of treatment is analyzed.
Measure: Mean (95% Confidence Interval); unit: Index score
Arm/Group | Amoxicillin | Azithromycin | Cotrimoxazole | Placebo
Number analyzed (Participants) | 31 | 31 | 31 | 31
Index score
  Baseline | 10.2 [8.8 to 11.5] | 8.8 [7.5 to 10.1] | 9.7 [8.2 to 11.2] | 9.6 [8.6 to 10.7]
  Post-treatment: number analyzed (Participants) | 27 | 30 | 29 | 29
  Post-treatment | 8.3 [7.0 to 9.6] | 6.6 [5.5 to 7.8] | 8.3 [6.9 to 9.7] | 9.8 [8.7 to 10.9]

12. Secondary Outcome: L2-norm Distance on Bacterial Reads (Nasopharyngeal)
Description: L2-norm distance on bacterial reads (nasopharyngeal)
Time Frame: Day 9
Population: Nasopharyngeal samples were not analyzed due to limited budget. these samples were collected but won't be analyzed.
Arm/Group | Amoxicillin Households | Azithromycin Households | Cotrimoxazole Households | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Macrolide Resistance Genes
Description: Prevalence of macrolide resistance genes measured using DNA-seq from rectal swabs.
Time Frame: 2 years
Population: The outcome is limited to children randomized to placebo in azithromycin households and to the placebo-treated child control in placebo households. A direct effect of antibiotics on the resistome was only observed among children receiving azithromycin compared with placebo; we were unable to process samples from the other study arms due to cost constraints.
  According to study design, only placebo treated children in these two arms were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Azithromycin Households: Eligible households that agreed to participate were randomized in a 1:1:1:1 fashion to a 5day course of amoxicillin, azithromycin, cotrimoxazole or placebo. Within each household, one child was randomized to the household's antibiotic assignment and one child to placebo. This group included children randomized to placebo in azithromycin households.
- Placebo Households: Eligible households that agreed to participate were randomized in a 1:1:1:1 fashion to a 5day course of amoxicillin, azithromycin, cotrimoxazole or placebo. Within each household, one child was randomized to the household's antibiotic assignment and one child to placebo. In placebo households, both children received placebo, and one child was randomly assigned to serve as the control for the antibiotic-treated child in the antibiotic households and one as the control for the placebo-treated child in the antibiotic households. This group included the placebo-treated child control in placebo households.
Arm/Group | Azithromycin Households | Placebo Households
Number analyzed (Participants) | 30 | 28
Participants | 12 | 9

14. Secondary Outcome: Alpha Diversity in the Intestinal Microbiome
Description: Alpha diversity in the intestinal microbiome using DNA-seq from rectal swabs
Time Frame: 2 years
Population: The intestinal microbiome in rectal swabs were not analyzed due to limited budget. these samples were collected but will not be analyzed
Arm/Group | Amoxicillin Households | Azithromycin Households | Cotrimoxazole Households | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: days 1-5
Description: On each day of treatment, caregivers were asked if the child had any symptoms since the previous day, including gastrointestinal symptoms, respiratory symptoms, a rash, or any other symptoms. Four days after the last treatment dose, caregivers were asked if their child had had three or more loose or watery stools over a 24-hour period, consistent with the WHO definition of diarrhea,21 and if the child currently had a cough or difficulty breathing.
Groups:
- Cotrimoxazole Households - Antibiotic: Households were randomized in a 1:1:1:1 fashion to a 5-day course of amoxicillin, azithromycin, cotrimoxazole, or placebo. Within each antibiotic household, one child was randomly assigned to receive placebo.
  Children will receive treatment everyday, once a day as is:
  Co-trimoxazole: 240 mg daily for Days 1-5
  Cotrimoxazole: Children in this arm will receive co-trimoxazole once a day. Cotrimoxazole: Children in this arm will receive co-trimoxazole once a day.
Arm/Group | Amoxicillin Households - Antibiotic | Amoxicillin Households - Placebo | Azithromycin Households - Antibiotic | Azithromycin Households - Placebo | Cotrimoxazole Households - Antibiotic | Cotrimoxazole Households - Placebo | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31 | 0/31 | 0/31 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31 | 0/31 | 0/31 | 0/60
Other Adverse Events (participants affected / at risk) | 5/31 | 0/31 | 3/31 | 5/31 | 3/31 | 3/31 | 7/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin Households - Antibiotic (N=31) | Amoxicillin Households - Placebo (N=31) | Azithromycin Households - Antibiotic (N=31) | Azithromycin Households - Placebo (N=31) | Cotrimoxazole Households - Antibiotic (N=31) | Cotrimoxazole Households - Placebo (N=31) | Placebo (N=60)
Vomiting, days 1-5 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea, days 1-5 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever, days 1-5 (General disorders) | 3 (3) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 3 (3)
Cough, Days 1-5 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Cough, Day 9 (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Diarrhea, days 1-5 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhea, day 9 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03187834/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03187834/SAP_001.pdf